CLINICAL TRIAL: NCT03164018
Title: Fampridine in MS Patients: A Cognition, Fatigue, Depression and Quality of Life Analysis
Acronym: FAMILY
Status: Completed | Type: Observational
Sponsor: Genesis Pharma CNS & Specialty (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GEN-FMP-001
Record Dates: First submitted 2017-03-29; First posted 2017-05-23 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fampridine — The non-interventional design allows the observation of patients in a broad range of settings reflecting routine clinical practice. All decisions on therapeutic or diagnostic procedures, treatments and management of the disease will be at the full discretion of the treating physician without interference by a sponsor or study protocol. All treatment decisions will follow the real-life treatment behavior.

SUMMARY:
Fampyra, a voltage-dependent potassium channel blocker, is indicated for the improvement of walking in adult patients with multiple sclerosis with walking disability (EDSS 4-7). The medicinal product has been authorized under a so-called "conditional approval" scheme. This means that further evidence on this medicinal product is awaited and this study aims to assess the effect of Fampyra, administered according to standard clinical practice, on cognition, fatigue and quality of life in patients with MS.

This clinical study is a multicenter, prospective, non-interventional, cohort study of MS patients receiving Fampyra in outpatient setting. Patients will be treated according to the local prescribing information of the study medication and routine medical practice in terms of visit frequency and types of assessments performed. The assignment of the patient to this therapeutic strategy is not decided in advance by the study protocol but falls within current practice and the prescription of Fampyra is clearly separated from the physician's decision to include the patient in the current study.

Since this is purely non-interventional study, primary data -which will be obtained prospectively during the study visits through patients' interview and patient reported outcomes or as performed per standard clinical practice- will mainly be employed.

DETAILED DESCRIPTION:
The study will take place in Greece. Investigator's decision to prescribe Fampyra (according to the indication for treatment as defined in the summary of product characteristics, SmPC and the current clinical practice), should precede entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old) with MS.
* Patient receiving Fampyra® for walking disability (EDSS 4-7).
* Patient receiving stable doses of any Disease Modifying Treatment (DMT) for at least 3 months prior to study entry.
* Patients will receive Fampyra® in line with the approved Summary of Product Characteristics (SmPC).
* Patients for whom the decision to prescribe therapy with Fampyra according to the locally approved product's summary of product characteristics (SmPC) has already been taken prior to their enrollment in the study and is clearly separated from the physician's decision to include the patient in the current study.
* Patients must have signed an informed consent document.
* Patients must be able to read, understand and complete the study specific questionnaires.

Exclusion Criteria:

* Pregnant or lactating woman.
* Patient with prior history or current presentation of seizure.
* Patient with mild, moderate or severe renal impairment (creatinine clearance < 80 ml/min).
* Concurrent treatment with other medicinal products containing fampridine (4-aminopyridine).
* Concomitant treatment with medicinal products that are inhibitors of Organic Transporter 2 (OCT2), e.g., cimetidine.
* Patients who have received more than 1 dose of fampridine at the time of enrollment into the study.
* Patients that meet any of the contraindications to the administration of the study drug according to the approved SmPC.
* Patients who currently receive treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with fampridine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the current clinical study is male and female patients with MS, aged ≥18 years, receiving Fampyra for walking disability according to standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in cognition measured with PASAT scale | Assessed at 2 weeks, 12 weeks and 24 weeks compared to Baseline (week 0).
  Correlated with the multidimensional Health Related Quality of Life in MS patients
Changes in depression measured with BDI-II scale | Assessed at 2 weeks, 12 weeks and 24 weeks compared to Baseline (week 0).
  Correlated with the multidimensional Health Related Quality of Life in MS patients
Changes in fatigue measured with MFIS scale | Assessed at 2 weeks, 12 weeks and 24 weeks compared to Baseline (week 0).
  Correlated with the multidimensional Health Related Quality of Life in MS patients
Changes in Quality of Life measured with MusiQoL scale | Assessed at 2 weeks, 12 weeks and 24 weeks compared to Baseline (week 0)
  Correlated with the multidimensional Health Related Quality of Life in MS patients
Changes in Quality of Life measured with MSIS-29 scale | Assessed at 2 weeks, 12 weeks and 24 weeks compared to Baseline (week 0)
  Correlated with the multidimensional Health Related Quality of Life in MS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Αiginitio hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mitsikostas DD, Doskas T, Gkatzonis S, Fakas N, Maltezou M, Papadopoulos D, Gourgioti R, Mitsias P. A Prospective, Observational, Cohort Study to Assess the Efficacy and Safety of Prolonged-Release Fampridine in Cognition, Fatigue, Depression, and Quality of Life in Multiple Sclerosis Patients: The FAMILY Study. Adv Ther. 2021 Mar;38(3):1536-1551. doi: 10.1007/s12325-020-01606-5. Epub 2021 Feb 2. PMID 33528792